CLINICAL TRIAL: NCT05736003
Title: Prolonged Versus Delayed Laparoscopic Cholecystectomy for Acute Cholecystitis: Time to Change the Concept - A Multicenter Randomized Controlled Trial
Brief Title: Prolonged Versus Delayed Laparoscopic Cholecystectomy for Acute Cholecystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Omar, MD, Associate professor of surgery, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVU/MED/SUR011/4/23/4/611
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged laparoscpic cholecystectomy (Experimental): Patients received laparoscopic cholecystectomy for acute cholecystitis after 27 hours of symptoms
  Interventions: Procedure: Laparoscopic cholecystectomy
- Delayed laparoscpic cholecystectomy (Active Comparator): Patients received laparoscopic cholecystectomy for acute cholecystitis after 6 weeks of symptoms
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Removal of gallbladder laparoscopically

SUMMARY:
Gallbladder stone affects 10-15% of the adult population, and about 15-25% of these patients presented with acute cholecystitis (AC). Laparoscopic cholecystectomy (LC) is considered the treatment of choice for patients with AC, and recent studies suggest that early laparoscopic cholecystectomy (ELC) is preferable. However, the optimal time for ELC in AC is still controversial.

Early laparoscopic cholecystectomy (ELC) was advised for patients presented within 72 hours, while conservative treatment and planned delayed laparoscopic cholecystectomy (DLC) after six weeks was recommended for patients presented after 72 hours. Surgeons almost always encounter patients with AC lasting more than 72 hours and these patients consistently refuse conservative treatment and postpone for the DLC.

DETAILED DESCRIPTION:
Gallbladder stone affects 10-15% of the adult population, and about 15-25% of these patients presented with acute cholecystitis (AC). Laparoscopic cholecystectomy (LC) is considered the treatment of choice for patients with AC, and recent studies suggest that early laparoscopic cholecystectomy (ELC) is preferable. However, the optimal time for ELC in AC is still controversial.

Early laparoscopic cholecystectomy (ELC) was advised for patients presented within 72 hours, while conservative treatment and planned delayed laparoscopic cholecystectomy (DLC) after six weeks was recommended for patients presented after 72 hours. ELC might be associated with a significant reduction in morbidity and mortality rates, comparable conversion rates, shorter hospital stays, lower costs, and higher patient satisfaction.

Surgeons almost always encounter patients with AC lasting more than 72 hours and these patients consistently refuse conservative treatment and postpone the DLC. Additionally, 15% of patients do not respond to the conservative treatment and still need an emergency cholecystectomy and another 25% of patients require re-hospitalization for recurrent attacks of AC and biliary colic, biliary pancreatitis, cholangitis, and calcular obstructive jaundice during the interval waiting for the DLC. Furthermore, DLC has a higher cost and is time-consuming.

Prolonged LC (PLC) for AC after 3 days from onset of symptoms was thought to be more technically difficult and dangerous because of altered anatomo-pathology where suppurative and subsequently necrotizing cholecystitis develops after edematous cholecystitis during the first 2 to 4 days of symptoms, and this may be associated with increased perioperative complications and conversion rate. On the contrary, others believed that hyperemia and edema may help the dissection. All the studies in the literature focus on the ELC and DLC with little data regarding the safety and feasibility of LC for acute cholecystitis beyond 72 hours of symptoms.

More clinical trials are needed for the optimal management of acute cholecystitis after 72 hours of symptoms. The aim of this study was to compare the clinical outcomes of prolonged and delayed LC in patients with acute cholecystitis more than 72 hours of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with acute cholecystitis beyond 72 hours of symptoms onset,
2. American Society of Anesthesiologists (ASA) scores I - III,
3. Aged 20-70 years,
4. Agreement to complete the study

Exclusion Criteria:

1. Gallbladder polyp,
2. common bile duct stones,
3. acute biliary pancreatitis,
4. cholangitis,
5. perforated cholecystitis,
6. biliary peritonitis,
7. pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Overall morbidity | 30 days
  The overall morbidity included failure of initial conservative treatment, emergency consultation, unplanned hospital readmission for recurrent attacks of AC or gallstone-related complications, subtotal cholecystectomy, and intra- and postoperative complications

SECONDARY OUTCOMES:
Morbidity | 30 days
  All intra and postoperative complications
Mortality | 30 days
  Death
Total length of hospital saty | 3 years
  Duration of hospitalization
Total Cost | 3 years
  The total cost includes the surgical and medical costs
Total antibiotic duration | 3 years
  Duration of antibiotic therapy
conversion rate | 3 years
  conversion from laparoscopic cholecystectomy to open cholecystectomy
Operative time | 3 hours
  duration from first trocar incision to last stitch
Lost days of work | 3 years
  Lost days of work

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Omar, M.D., Principal Investigator — General Surgery Department, Faculty of Medicine, South Valley University
Locations (1):
- Mohammed Ahmed Omar, Luxor, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For 1 year
Access Criteria: After publication